CLINICAL TRIAL: NCT06268457
Title: Chemioembolizzazione Arteriosa Per il Trattamento Della Fibromatosi Desmoide: Studio Osservazionale Prospettico
Brief Title: Arterial Chemoembolization for the Treatment of Desmoid Fibromatosis
Acronym: Embodesmo
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: CE-AVEC 789/2023/Oss/IOR
Record Dates: First submitted 2024-02-08; First posted 2024-02-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Desmoid
Keywords: Chemoembolization
MeSH Terms: conditions — Desmoid Tumors | interventions — Doxorubicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Performed chemoembolization
  Interventions: Procedure: Chemoembolization with Doxorubicin

INTERVENTIONS:
Procedure: Chemoembolization with Doxorubicin — * Identification of the main vessels afferent to the metastasis to be treated.
  * Selective and super-selective catheterization of pathological arterial branches, responsible for the blood supply to the neoplasm, through the use of micro-catheters.
  * Injection of embolizing material (hydrogel microspheres with doxorubicin)
  * Control of technical success: the embolization will be followed by diagnostic arteriography that will evaluate the success of the procedure (occlusion of more than 90 percent of the pathologic vasculature).

SUMMARY:
Desmoid fibromatoses are rare (1-2 cases/million per year) and locally aggressive mesenchymal tumors. For asymptomatic disease, current guidelines suggest an initial period of active surveillance.

The current scientific evidence regarding the efficacy and safety of the treatment of desmoid fibromatosis by arterial embolization is constituted by several retrospective and prospective studies. Embolization of desmoid tumors alone, without chemotherapy, on the contrary, has been shown to be inefficient. Using Doxorubicin in desmoid fibromatosis is effective but associated with systemic toxicity. Consequently, this drug is reserved for symptomatic, nonresponsive, rapidly growing or life-threatening tumors. The intrinsic hypervascularity of desmoid tissue can be exploited as a conduit to achieve local distribution of Doxorubicin by navigation of a catheter endovascular.

DETAILED DESCRIPTION:
Desmoid fibromatoses are rare (1-2 cases/million per year) and locally aggressive, characterized histologically by monoclonal myoblasts present in abundant stromal tissue.The current therapeutic strategy has abandoned primary resection, as recurrences after resection are common and often their phenotype is more infiltrative. Nonsurgical approaches remain suboptimal. For asymptomatic disease, current guidelines suggest an initial period of active surveillance.

The current scientific evidence regarding the efficacy and safety of the treatment of desmoid fibromatosis by arterial embolization is constituted by several retrospective and prospective studies. These studies report promising results through the use of chemoembolization, that is, arterial embolization using particles loaded with chemotherapy. Embolization of desmoid tumors alone, without chemotherapy, on the contrary, has been shown to be inefficient. Doxorubicin is routinely used in the treatment of soft tissue sarcomas and other mesenchymal malignancies. Its use against desmoid fibromatosis is effective but associated with hematologic, gastrointestinal, and cardiac toxicity. Consequently, this drug is reserved for symptomatic, nonresponsive, rapidly growing or life-threatening tumors. The intrinsic hypervascularity of desmoid tissue can be exploited as a conduit to achieve local distribution of Doxorubicin by navigation of a catheter endovascular. Doxorubicin contains a protonated amine group which can establish an ionic bond with the sulfonate present on the surface of microbeads of hydrogel, ensuring embolization and elution of the drug. This process allows high concentrations of Doxorubicin in the target tissue and low concentrations in the systemic circulation.

ELIGIBILITY:
Inclusion Criteria:

* FIbromatosis demsoid symptomatic and in active phase (documented growth at last follow-ups)
* Patients who are not candidates for surgery or cryoablation

Exclusion Criteria:

* Patients with life expectancy <3 months or severely impaired status functional status (ASA 4)
* Patients with fibromatosis not in active phase, documented clinically and by investigations imaging (MRI, CT)
* Patients with coagulation deficiency or plateletopenic disease
* Patients with documented active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by desmoid fibromatoses eligible to be treated with chemoembolization with Doxorubicin
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Volume reduction in cm | 1 year
  Reduction of the lesion evaluated with MRI, measuring the diameter of the lesion in cm.
Reduction of pain (VAS score) | 1 year
  Clinical assessment regarding pain by Visual Analogue Scale (VAS) score (0-100 mm), in which 0 represents no pain, and 100 represents maximum pain imaginable.
Reduction of antalgic therapy (mg) | 1 year
  Mean reduction in the use of pain medications evaluated in mg of active ingredient taken daily before the treatment and at follow-up.

SECONDARY OUTCOMES:
Improvement in quality of life (EORTC QLQ-C15-PAL questionnaire) | 1 year
  Clinical assessment regarding quality of life by EORTC QLQ-C15-PAL questionnaire. The questionnaire consists of several scales, covering different aspects related to palliation. The maximum and minimum scores for each scale of the questionnaire can range from 0 to 100. The interpretation of scores depends on the specific scale in the questionnaire, and a higher value may indicate either greater negative impact (e.g., more symptoms or more suffering) or greater positive impact (e.g., better quality of life or less symptomatology). The overall assessment requires a detailed analysis of individual scores and related scales.
Improvement in quality of life (EORTC QLQ - BM22) | 1 year
  Clinical assessment regarding quality of life by EORTC QLQ - BM22 questionnaire. The questionnaire consists of several scales, covering different aspects related to palliation. The maximum and minimum scores for each scale of the questionnaire can range from 0 to 100. The interpretation of scores depends on the specific scale in the questionnaire, and a higher value may indicate either greater negative impact (e.g., more symptoms or more suffering) or greater positive impact (e.g., better quality of life or less symptomatology). The overall assessment requires a detailed analysis of individual scores and related scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy